CLINICAL TRIAL: NCT06919926
Title: A Randomized, Within-subject, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of AGB101 (Low-dose Levetiracetam, 220 mg, Extended Release Tablet) for the Treatment of Hippocampal Overactivity in the Elderly
Brief Title: Clinical Trial Evaluating the Efficacy of AGB101 for Reducing Hippocampal Overactivity in Older Adults
Acronym: AGB101-CN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: AgeneBio (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00437850; 5R01AG061091 (NIH)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hippocampal Overactivity; Dementia
MeSH Terms: conditions — Dementia | interventions — Levetiracetam; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AGB101 first, then placebo (Experimental): AGB101 (low-dose levetiracetam, 220 mg, extended release tablet) once daily for 2 weeks, washout (4 weeks), then placebo capsule once daily for 2 weeks.
  Interventions: Drug: AGB101; Drug: Placebo
- placebo first, then AGB101 (Experimental): Placebo capsule once daily for 2 weeks, washout (4 weeks), then AGB101 (low-dose levetiracetam, 220 mg, extended release tablet) once daily for 2 weeks.
  Interventions: Drug: AGB101; Drug: Placebo

INTERVENTIONS:
Drug: AGB101 — low-dose levetiracetam, 220 mg, extended release tablet
  Other Names: levetiracetam
Drug: Placebo — placebo capsule
  Other Names: sugar pill

SUMMARY:
This randomized, crossover, placebo controlled clinical study will assess the efficacy and safety of a slow release form of levetiracetam (AGB101) in the treatment of cognitively normal adults by measuring change in several imaging measures over the course of a two week treatment period.

DETAILED DESCRIPTION:
In clinical studies, the magnitude of hippocampal over-activity longitudinally predicts subsequent cognitive decline/conversion to dementia, and hippocampal over-activity in subjects with mild cognitive impairment (MCI) due to Alzheimer's disease (AD) is significantly correlated with the extent of neuronal injury affecting AD-specific regions of the brain. A previous study reported a significant correlation between greater hippocampal activation (fMRI) and more pronounced medial temporal lobe (MTL) atrophy (cortical thinning) indicative of AD-related neurodegeneration in subjects with MCI due to AD with a Clinical Dementia Rating (CDR) score of 0.5 selected by Alzheimer's Disease Neuroimaging Initiative (ADNI)-1 criteria. This supports a therapeutic rationale to reduce over-activity in order to slow or prevent neuronal injury.

Modest hippocampal over-activity has also been observed in preclinical (asymptomatic) conditions in older adults. In previous studies, older adults showed increased hippocampal activation compared to young adults in the context of cognitive performance within the normal range for the participant's age. These findings suggest that hippocampal over-activity may be an opportunity for early intervention examining whether treatment of hippocampal over-activity early in the progression confers benefit to older adults at risk for AD dementia. The current study aims to test this hypothesis in cognitively normal subjects between the ages of 50 and 80.

ELIGIBILITY:
Subjects must meet all of the following inclusion criteria at screening:

1. Subjects between 50 and 80 years old (inclusive) in good general health:

   1. Willing and able to consent and participate for the duration of the study.
   2. Have eighth-grade education or good work history sufficient to exclude mental retardation.
   3. Have visual and auditory acuity adequate for neuropsychological testing.
   4. Have proficient fluency of the native local language to participate in all the neuropsychological test assessments.
2. Have a study partner who has sufficient contact (≥ 2 hours per week) with the subject and can provide assessments of any changes and an independent evaluation of the subject's functioning.
3. Have normal cognition as defined by the following criteria:

   1. Mini-Mental State Examination (MMSE) scores between 27 and 30 (inclusive; exceptions may be made for subjects with < 12 years of education at the discretion of the investigator)
   2. No memory complaint reported by the subject or his/her study partner.
   3. Evidence of normal memory function documented by a normal score on the Buschke Selective Reminding Test Immediate and Delayed Recall or equivalent test.
   4. A Clinical Dementia Rating Scale (CDR) global score of 0 with a memory box score of 0.
4. Antidepressants must be at a stable dose for 1 month prior to screening and expected to remain stable throughout the study.
5. Willing and able to undergo repeated MRI scans (3 Tesla) with no contraindications to MRI.
6. Willing to allow collection of blood for apolipoprotein E (ApoE) genotyping and banking.
7. Willing and able to undergo a Tau positron emission tomography (PET) scan with 18F MK-6240 tracer.
8. If female participant or partner/spouse is of childbearing age, participant and/or partner must be willing to use an effective contraception for duration of the study and for 4 days after it. For women, effective contraception may be hormonal; for men, a condom.

Exclusion Criteria:

* Subjects must not meet any of the following exclusion criteria at screening:

  1. Use of anticonvulsant or anticoagulant medications within 1 month prior to the baseline visit.
  2. Participation in a therapeutic clinical study for any medical or psychiatric indications within 1 month of the screening visit, or at any time during the study. Subjects must understand that participants may only enroll in this clinical study once; participants may not enroll in any other clinical study while participating in the current study, and participants may not participate in a clinical study of a drug, biologic, therapeutic device, or medical food, in which the last dose/administration was received within 1 month prior to screening.
  3. History of hypersensitivity or lack of tolerability to AGB101 (levetiracetam).
  4. Severe renal impairment (creatinine clearance of < 30 mL/minute) or undergoing hemodialysis.
  5. Any significant neurological disease such as Parkinson's disease, Alzheimer's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder (lifetime history; infant febrile seizures are not exclusionary), subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits, or known structural brain abnormalities, that in the opinion of the investigator might interfere with the conduct of the study.
  6. Diagnosis of major depression within the last 3 years or prior diagnosis of schizophrenia, bipolar disorder or other psychotic disorder.
  7. Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, or body that constitute a contraindication to having an MRI scan.
  8. History of alcohol or substance abuse or dependence within the past 3 years (DSM-5 criteria).
  9. Any significant systemic illness or unstable medical condition that could lead to difficulty in complying with the protocol requirements.
  10. Any unstable medical condition that is likely to require new medical or surgical treatment during the course of the study and where such treatments might affect the collection of efficacy data.
  11. Current suicidal ideation.
  12. Female subjects must not be pregnant or lactating.
  13. Any other reason, which in the opinion of the investigator would confound proper interpretation of the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in hippocampal overactivity as measured by fMRI (functional Magnetic Resonance Imaging) | Week 2, Week 8
  The primary efficacy evaluation is confirmation of target engagement demonstrated by reduction in hippocampal overactivity comparing the end of the active treatment period compared to the end of the placebo treatment condition as measured by task-based functional magnetic resonance imaging.

SECONDARY OUTCOMES:
Change in functional connectivity measures as measured by fMRI (functional Magnetic Resonance Imaging) | Week 2, Week 8
  Functional connectivity measures comparing the end of the active treatment period to the end of the placebo treatment condition as measured by resting state fMRI (functional Magnetic Resonance Imaging).

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Bakker, Ph.D., Study Director — Johns Hopkins University; Marilyn Albert, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yassa MA, Lacy JW, Stark SM, Albert MS, Gallagher M, Stark CE. Pattern separation deficits associated with increased hippocampal CA3 and dentate gyrus activity in nondemented older adults. Hippocampus. 2011 Sep;21(9):968-79. doi: 10.1002/hipo.20808. Epub 2010 May 20. PMID 20865732
- [Background] O'Brien JL, O'Keefe KM, LaViolette PS, DeLuca AN, Blacker D, Dickerson BC, Sperling RA. Longitudinal fMRI in elderly reveals loss of hippocampal activation with clinical decline. Neurology. 2010 Jun 15;74(24):1969-76. doi: 10.1212/WNL.0b013e3181e3966e. Epub 2010 May 12. PMID 20463288
- [Background] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Background] Dickerson BC, Salat DH, Greve DN, Chua EF, Rand-Giovannetti E, Rentz DM, Bertram L, Mullin K, Tanzi RE, Blacker D, Albert MS, Sperling RA. Increased hippocampal activation in mild cognitive impairment compared to normal aging and AD. Neurology. 2005 Aug 9;65(3):404-11. doi: 10.1212/01.wnl.0000171450.97464.49. PMID 16087905
- [Background] Miller SL, Fenstermacher E, Bates J, Blacker D, Sperling RA, Dickerson BC. Hippocampal activation in adults with mild cognitive impairment predicts subsequent cognitive decline. J Neurol Neurosurg Psychiatry. 2008 Jun;79(6):630-5. doi: 10.1136/jnnp.2007.124149. Epub 2007 Sep 10. PMID 17846109